CLINICAL TRIAL: NCT01924637
Title: A Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of FIAsp in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3889; 2011-000941-19 (EudraCT Number); U1111-1119-5708 (Other: WHO)
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIASP (Experimental): Each treatment period consists of 1 dosing visit during which the subject will receive a single dose of either insulin aspart or FIAsp at a predefined fixed dose level (in random sequence) in connection to intake of a standardised meal.
  Interventions: Drug: Faster-acting insulin aspart
- NovoRapid® (Active Comparator): Each treatment period consists of 1 dosing visit during which the subject will receive a single dose of either insulin aspart or FIAsp at a predefined fixed dose level (in random sequence) in connection to intake of a standardised meal.
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — A single dose will be administered subcutaneously (under the skin) in the abdomen.
  Each subject will be allocated to two treatment periods separated by a wash-out period of 3-12 days.
  Arms: FIASP
Drug: insulin aspart — A single dose will be administered subcutaneously (under the skin)) in the abdomen.
  Each subject will be allocated to two treatment periods separated by a wash-out period of 3-12 days.
  Arms: NovoRapid®

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetic (the exposure of the trial drug in the body) and pharmacodynamic (the effect of the investigated drug on the body) properties of FIAsp (faster-acting insulin aspart) in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.5-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mean change in plasma glucose concentration | From 0-2 hours after administration

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 1 hour
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Background] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. Faster Onset and Greater Early Exposure and Glucose-Lowering Effect with Faster-Acting Insulin Aspart vs. Insulin Aspart: A Pooled Analysis in Subjects with Type 1 Diabetes. Diabetes. 2016; Suppl. 1: A239. doi:10.2337/db16-861-1374 http://dx.doi.org/10.2337/db16-861-1374
- [Derived] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. A Pooled Analysis of Clinical Pharmacology Trials Investigating the Pharmacokinetic and Pharmacodynamic Characteristics of Fast-Acting Insulin Aspart in Adults with Type 1 Diabetes. Clin Pharmacokinet. 2017 May;56(5):551-559. doi: 10.1007/s40262-017-0514-8. PMID 28205039
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com